CLINICAL TRIAL: NCT04525625
Title: Risk Factors for Acute Kidney Injury in Critically Ill Patients With Acute-on-Chronic Liver Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institutul Clinic Fundeni (Other)
Responsible Party: Principal Investigator, Popescu Mihai, clinical professor, Institutul Clinic Fundeni
Other Study IDs: AKI-ACLF
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Acute Kidney Injury; Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute Kidney Injury; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute kidney injury (AKI) is one of the most important factors associated with increased mortality in patients with acute-on-chronic liver failure (AoCLF). Early identification and treatment of this subgroup of patients may improve survival and decrease ICU length of stay. As kidney ischemia is one of the main mechanisms responsible for AKI in AoCLF, an increase in urinary to arterial partial pressure of oxygen may help in the early diagnosis of renal failure. For this arterial and urinary oxygen pressure will be measured at ICU admission, on day 1 and day 3 of ICU stay. Diagnosis of AKI within the first 28 days after ICU admission will be recorded

ELIGIBILITY:
Inclusion Criteria:

- patients admitted to the ICU for acute-on-chronic liver failure

Exclusion Criteria:

* pre-existing renal disease
* urine output<200 mL/day
* death within the first 24 hours after ICU admission
* emergency liver transplantation within the follow-up period (28 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted to a general ICU for ACLF who fall into the inclusion and exclusion criteria. Standard treatment will be applied to all patients and no supplemental intervention is required for the present study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
AKI | 28 days after ICU admission
  incidence (%) of AKI in patients with AoCLF as defined by Acute Kidney Injury Network guidelines

SECONDARY OUTCOMES:
arterial to urinary oxygen gradient | ICU admission, ICU day 1 and ICU dy 3
  mathematical difference in oxygen partial pressure between arterial blood and urine (mmHg) in patients with AKI compared to patients without AKI
mortality | 28-days
  28-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Dana Tomescu, Prof, Study Chair — Fundeni Clinical Institute
Locations (1):
- Popescu Mihai, Bucharest, Romania